CLINICAL TRIAL: NCT02516371
Title: Lymphocytes Subpopulation and Its Relevance With Tumor Grade and Prognosis in Cancer Patients
Brief Title: Lymphocytes Subpopulation in Cancer Patients
Acronym: CaLym
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: DERSHENG SUN (Other)
Responsible Party: Sponsor-Investigator, DERSHENG SUN, Clinical assistant professor, The Catholic University of Korea
Organization: The Catholic University of Korea (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UC15OISI0093
Record Dates: First submitted 2015-08-01; First posted 2015-08-05 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Lymphocyte Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lymphocytes (Other): To evaluate the subpopulation of lymphocytes in cancer patients
  Interventions: Other: lymphocyte

INTERVENTIONS:
Other: lymphocyte — To evaluate the subpopulation of lymphocytes in cancer patients
  Other Names: subpopulation of lymphocytes in cancer patients

SUMMARY:
This study aims to exam the subpopulation of lymphocytes and evaluate the clinico-pathologic correlations.

DETAILED DESCRIPTION:
The host's inflammatory response in the tumor microenvironment could effect cancer progression and prognosis. As components of systemic inflammatory response, lymphocytes, neutrophils, and platelets are being recognised to have an important role in carcinogenesis and tumor progression. To date, a number of peripheral blood-derived inflammation-based scores such as the neutrophil-lymphocyte ratio (NLR), platelet- lymphocyte ratio (PLR) and so on have been proposed as prognostic markers in numerous types of cancers. But, very little is known of their impact in subpopulation of lymphocytes. The investigators try to evaluate the activity of lymphocytes in peripheral blood and find out the relationship among clinical prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. cancer patients of Uijeongbu St. Mary's Hospital
2. never treated with chemotherapy
3. Age between 20~80 years-

Exclusion Criteria:

1. treated with chemotherapy before
2. No informed consent form

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
response rate after cancer treatment with chemotherapy | 6 months after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Ho Ko, MD, PhD, Principal Investigator — Uijeongbu St. Mary's Hospital, The Catholic University of Korea
Locations (1):
- Uijeongbu St. Mary's hospital, the Catholic university of Korea, Uijeongbu-si, Gyounggido, South Korea